CLINICAL TRIAL: NCT02123030
Title: A Micro/Nano Device for Exhaled Breath Analysis
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Xiao-An Fu, Assistant Professor, University of Louisville
Other Study IDs: 10.0642
Record Dates: First submitted 2014-04-22; First posted 2014-04-25 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer; Pulmonary Disease
Keywords: Lung cancer; pulmonary disease
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breathe samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental: patients with pulmonary disease; and, patients with known or suspected lung or other cancers
- Control: healthy subjects (for example, family members of the patient or graduate students

SUMMARY:
Use of a microfabricated silicon device to concentrate ultra trace volatile organic compounds (VOCs) in human exhaled breath for quantitative analysis of VOCs.

DETAILED DESCRIPTION:
Will use Fourier Transform Mass Spectrometry (FT-MS) and Gas Chromatography-Mass Spectrometry (GC-MS) to analyze concentrated VOCs. The purpose of this study is to search for disease-related markers in the breath in subjects with known or suspected lung or other cancer, or pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* For controlled (healthy) subjects - we are seeking persons who do not have a known history of cancer or pulmonary disease.
* Both smokers and nonsmokers are invited to participate as control subjects.
* For experimental subjects, we are seeking persons with pulmonary disease but no known history of cancer, as identified by the investigators during routine clinic or office visits.
* Additionally for experimental subjects, we are seeking persons with known or suspected lung or other cancers, as identified by the investigators during routine clinic or office visits.

Exclusion Criteria:

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those fitting inclusionary criteria between 20 and 85 years of age, with or without history of pulmonary disease or cancer.
Sampling Method: Non-Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Detection of disease related markers (biomarkers) from concentrated volatile organic compounds in breath samples | 1 day (After sample collection)
  The concentrated volatile organic compounds in exhaled breath samples will be analyzed by statistical software for search for disease related markers (biomarkers).

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-An Fu, PhD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center-University of Louisville, Louisville, Kentucky, United States